CLINICAL TRIAL: NCT01367041
Title: Effect of Hip Bone Mineral Density / Content on Vibration-Induced Hip Adductors Muscle Electrical Activity in Postmenopausal Women
Brief Title: Effect of Bone on Vibration-Induced Muscle Electrical Activity
Acronym: PMO-WBV-sEMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Karacan, Chief of Physical Med & Rehab Clinic, Bagcilar Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BEAH FTR-3; NCT00961545 (obsolete NCT alias)
Record Dates: First submitted 2011-04-06; First posted 2011-06-06 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Osteoporosis
Keywords: bone; muscle electrical activity; whole-body vibration
MeSH Terms: conditions — Osteoporosis | interventions — Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone loss (Experimental): Postmenopausal women with osteoporosis, whole body vibration will be applied at 40 Hz, 2mm amplitude, 30+30s
  Interventions: Procedure: vibration
- Normal (Experimental): Postmenopausal women without osteoporosis, whole body vibration will be applied at 40 Hz, 2mm amplitude, 30+30s
  Interventions: Procedure: vibration

INTERVENTIONS:
Procedure: vibration — Vibration frequency: 40 Hz, duration: 30+30 s, 2mm amplitude

SUMMARY:
The aim of this study is to investigate effects of femur exposed to vibration on the rest muscle electrical activity of hip adductors in cases with postmenopausal osteoporosis.

Among patients who will be admitted to the investigators clinic for out-patients and whose bone densitometric measurement will be made with a prediagnosis postmenopausal osteoporosis, a total of 80 voluntaries [40 having postmenopausal osteoporosis (femur neck or total hip T score < -2.0) and 40 Controls (Hip and lumbar bone mineral density normal)] are planned to include in this study.

After the left hip bone mineral density (BMD) and BMC is measured in all cases, whole body vibration will be applied in PMO groups and Controls. The rest muscle electrical activity of left hip muscles will be evaluated at pre-treatment, post-treatment and, during treatment in patients with PMO and then their data will be compared with Controls data.

Plasma sclerostin level will be measured before and 10th minute after vibration.

Cases will stand on vibration plate. WBV will be applied at a frequency of 40 Hz and amplitude of 2 mm for 30 + 30 seconds. WBV will be applied one session only. The left hip BMD and BMC will be evaluated by bone densitometer (Norland).

The rest muscle electrical activity of hip adductor muscles at rest will be measured by PowerLab (data acquisition system, ADInstruments, Australia) device.

This project is planed to be completed in 3 months.

DETAILED DESCRIPTION:
It is usually reported that there is a parallelism between changes in the bone structure and function and the muscle structure and function. Sarcopenia is frequently observed in osteoporotic patients. Bone formation increases or bone resorption decreases with exercise.

One of the most important functions of bone bear mechanical loads include body weight. Bone must be strong enough to resist the mechanical loading. Mechanisms need to protect bone when bone is subject to excessive mechanical loading. These mechanisms may mainly focus on strengthening the bone and/or changing vectorial properties of mechanical loading applied bone.

The vectorial properties of mechanical loading applied bone may be controlled by muscle contractions. Bone contains wide mechanoreceptor net constructed by osteocytes. So,distribution of the mechanical loading on bone cross-sectional area is possible to perceive. It may be also possible that inappropriate distribution of mechanical loading on bone crosssectional area is optimized by muscle contractions. To get this regulation, there should be a mechanism that muscle activity is controlled by central nervous system based on mechanical loading distribution on bone cross-sectional area. The investigators previously showed that bone can regulate muscle activity, based on its bone mineral density. According to this study result, it can be suggested there may exist a mechanism that bone sensing mechanical stimuli can send the signals to central nervous system and neuronally regulate muscle activity (bone myo-regulation reflex). (It is also well known that load-induced adaptive bone formation is neuronally regulated. Taken together, a general mechanism, bone reflex, may be defined that bone subjected to loading can neuronally regulate bone formation and muscle activity) Vibration has a strong osteogenic effect. Vibration-induced bone formation is neuronally regulated. Vibration can also effectively enhance muscle strength and power. Previous studies have shown that vibration increases muscle electromyographic (EMG) activity. It has been showed that bone has an effect on the increase in muscle EMG activity caused by vibration in healthy young adults in a study. In this study, it was reported that vibrations-induced increases in muscle electrical activity of flexor carpi radialis (FCR) was related to ultradistal radius bone mineral content (BMC) and the FCR H-reflex was suppressed or depressed during vibration. This findings were reported to support the assumption that the bone exposed to cyclic mechanical loading may neuronally regulate muscle activity.

The aim of this study is to investigate effects of femur exposed to vibration on the rest muscle electrical activity of hip adductors in cases with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with osteoporosis(femur neck or total hip T score<-2) or postmenopausal women without osteoporosis (normal femur and lumbar bone mineral density)
* women with ages varying between 45 and 65 years
* right handed women

Exclusion Criteria:

* secondary osteoporosis, fracture history
* early menopause
* osteopenia (-2 < femur neck or total hip T score < 1)
* neuropathy (central or peripheral)
* muscle, tendon, joint, vascular, dermatologic disease in lower extremity
* postural abnormality (scoliosis, kyphosis,short leg etc)
* systemic diseases (severe hypertension, coronary heart disease, etc)
* endocrine-metabolic bone diseases[paget, osteomalacia]
* medication that could affect the musculoskeletal system
* obesity (BMI >30 kg/m2 or body weight>80kg)
* professional sportswoman
* female doing regular sports activities
* non-cooperative subject
* vertigo

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Vibration-induced muscle electrical activity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)